CLINICAL TRIAL: NCT02498301
Title: A Randomized, Placebo-Controlled, Double-Blind, Clinical Trial Evaluating Two Dose Regimens of Rifaximin (550 mg Daily or 550 mg Twice Daily) for Chemoprophylaxis Against Travelers' Diarrhea (TD) Among Active Duty Deployed U.S. and British Military Personnel
Brief Title: Trial Evaluating Chemoprophylaxis Against Travelers' Diarrhea - Prevent TD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Naval Medical Research Center (U.S. Federal Agency); Ministry of Defence, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IDCRP-080
Record Dates: First submitted 2015-07-06; First posted 2015-07-15 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2021-11

CONDITIONS: Travelers' Diarrhea; Functional Bowel Disorders; Reactive Arthritis
Keywords: travelers' diarrhea; military; enteric illness; gastrointestinal
MeSH Terms: conditions — Arthritis, Reactive | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rifaximin 550 mg once/day (Experimental): rifaximin, 550 mg, once daily, by mouth
  Interventions: Drug: Rifaximin
- Rifaximin 550 mg twice/day (Experimental): rifaximin, 550 mg, twice daily, by mouth
  Interventions: Drug: Rifaximin; Drug: Placebo
- Placebo (Placebo Comparator): Placebo pills, twice daily, by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Rifaximin will be provided to subjects either daily with placebo, or twice daily depending on which of the two experimental arms they are randomized to
  Other Names: Xifaxan
  Arms: Rifaximin 550 mg once/day; Rifaximin 550 mg twice/day
Drug: Placebo — Placebo will be administered twice daily or once daily with rifaximin depending on which experimental arm they are randomized to
  Arms: Placebo; Rifaximin 550 mg twice/day

SUMMARY:
The purpose of this study is to develop evidence on the relative efficacy of 2 rifaximin chemoprophylaxis regimens for the prevention of Travelers' Diarrhea (TD) in a deployed setting. An additional purpose is to explore the effect of chemoprophylaxis on microbial flora and antimicrobial resistance, and obtain parameter estimates to inform a cost-effectiveness model of chemoprophylaxis in prevention of TD. Information from this study will be used to develop management guidelines for the prevention of TD among deployed (United States (US) and United Kingdom (UK) military personnel.

The study will be a multi-site, randomized, placebo-controlled, double-blind, clinical trial among deployed military personnel. The study will test 2 TD chemoprophylaxis regimens (once daily versus twice daily) of the same antibiotic, rifaximin, compared to a placebo.

For the proposed chemoprophylaxis study described herein, cohorts of military personnel (US and UK) deploying/traveling overseas will be recruited prior to travel to participate and will undergo enrollment procedures as outlined in study appendices. Subjects who are eligible and agree to participate will be randomized to receive one of 3 regimens: (1) rifaximin 550 mg daily; (2) rifaximin 550 mg twice a day; or (3) placebo, to be taken while deployed. Chemoprophylaxis will be maintained for duration of travel or a predetermined period of up to 6 weeks and at least 2 weeks, which may include a period of up to 5 days of use after return to COO for deployments less than 6 weeks in duration. Clinical and laboratory data will be obtained before, during if available and after deployment/chemoprophylaxis.

DETAILED DESCRIPTION:
The primary efficacy outcome will be assessed by review of the symptom memory aid (TravMil diary). Subjects will follow a symptom memory aid from the onset of a disease episode and record relevant symptomatology (date/time and number of diarrheal episodes, associated symptoms such as fever, vomiting, nausea, bloody stools and cramps, severity of symptoms, functional activity). Use of antibiotics and/or Imodium (loperamide) for each episode will also be recorded). An additional memory aid to capture occurrence of solicited adverse events, use of new prescription medications, as well as adherence to study medication regimen will be utilized by subjects during deployment and returned (or re-created with study personnel if lost or incomplete) at follow-up Memory aid data will be actively sought from all subjects via required in-person follow-up.

Secondary efficacy outcomes will also largely be derived from the self-report of subjects via use of the memory aid data. Secondary safety evaluation will be performed at the end of study visit based on history obtained from the subject regarding medical treatment requiring events while deployed.

Individuals will be enrolled prior to travel/deployment. At the time of enrollment they will undergo eligibility criteria review, informed consent process, baseline assessment (demographics, medical history, others), sample collection (blood and stool), and blinded randomization into a study arm.

Episodes of diarrhea are expected to occur while on study drug. Subjects will be instructed and expected to seek care for these episodes from medical assets available to them at COD.

Subjects will be instructed to discontinue study drug if they develop diarrhea and are given antibiotic therapy. It is not expected that study drug will impact the choice or effectiveness of antibiotics used to treat travelers' diarrhea. Some subjects will be eligible to restart (only once restart) study drug once they are cured of a travelers' diarrhea episode. See US and UK addenda for details.

The end of prophylaxis is defined as the +/- 96hr period from cessation of prophylaxis due to (A) the subject completing maximal period of prophylaxis but remains deployed, or (B) being re-deployed and returns to mainland/COO. During this end of prophylaxis period, subjects may be seen by study personnel and perform an end of prophylaxis visit.

The post-deployment period is defined as the return to COO through 8 weeks from return. A post-deployment visit, in the COO will be planned for all subjects enrolled in the study and will occur as soon as it can be scheduled.

All subjects will be asked to complete a baseline questionnaire on day of enrollment and complete web-based surveys during the follow-up period. Subjects will be emailed the survey link at 3 and 6 months post-return to COO. The survey will assess for several types of functional bowel disorders and symptoms of ReA using standardized questions and definitions and questions and will use disease activity scales to assess impact on daily life.

A sample of blood will be collected up to 2 times as part of participation in this study. The samples will be collected, processed and stored until transported at a later date to central lab for testing of acute and convalescent titers directed against bacterial and viral enteropathogens. Samples will also be used for biomarker evaluation and support of exploratory objectives.

Stool samples will be used for exploratory microbiological analyses to assess etiology of diarrhea by pathogen, antibiotic susceptibility of enteropathogens, and evaluation of impact of rifaximin on the microbiome. Serum will be utilized to attempt to determine seroconversion status for pathogens not identified during stool analysis.

ELIGIBILITY:
Inclusion Criteria:

1. An Institutional Review Board (IRB) / Ethics Committee (EC)-approved informed consent form is signed and dated.
2. Subject is at least 18 years of age
3. Subject's duration of prophylaxis will be least 2 weeks.
4. Subject is capable of and willing to comply with all study procedures and available for the end of study visits and sample collection at COO (within 6 months from start of prophylaxis).
5. Women: Non-nursing and negative urine/serum pregnancy test with understanding (through informed consent process) to avoid pregnancy while on study drug. Sole reliance on oral contraceptives (OCPs) for birth control will not be recommended (see section 6.3.2.1.) Should an individual have a documented surgical sterilization in her medical record, a pregnancy test will not be required. If a volunteer becomes pregnant during the study, the principal investigator will notify the study research monitor and the IRBs. The pregnancy outcome will be followed per IRB and other regulatory requirements for US and UK personnel.
6. (For US Personnel Only). Have consented to participate in TravMil protocol.

Exclusion Criteria:

1. Subject received any systemic or gastrointestinal antibiotic in the 7 days prior to enrollment (except anti-malarial prophylaxis agents).
2. Subject has hypersensitivity or allergy to rifaximin or rifampicin.
3. Subject has acute diarrhea within 7 days prior to enrollment
4. Subject has a concomitant disease or condition that could interfere with, or for which treatment could interfere with, the conduct of the study, or could in the opinion of the investigator increase the risk of AEs during the subject's participation in the study
5. Subject is currently taking or plans to take during deployment at least one of the following medications: theophylline or warfarin (Coumadin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2015-11-10 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy - Risk of travelers diarrhea during chemoprophylaxis as measured by self-report via use of a memory aid | 24hr

SECONDARY OUTCOMES:
Efficacy as determined by use of a symptom memory aid. | For a duration of prophylaxis which will be on average 3-4 weeks or a maximum of 6 weeks
  Proportion of subjects in each treatment group with TD, with mild diarrhea, with TD associated with isolation of a pathogen and pathogen type, total diarrhea days, work days and performance loss due to diarrhea, comparison of incidence of TD
Solicited adverse events as collected from the subject and using a memory aid | For the duration of prophylaxis which will be on average 3-4 weeks or a maximum of 6 weeks.
  Solicited adverse events will be collected by use of a memory aid which will be reviewed at the last clinic visit, on average within 4 months from study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Ramiro Gutierrez, MD, Principal Investigator — Naval Medical Research Center
Locations (6):
- United States (5):
  - Naval Medical Center San Diego, San Diego, California
  - Tripler Army Medical Center/Schofield Barracks, Honolulu, Hawaii
  - Naval Hospital Camp Lejeune, Marine Corps Base Camp Lejeune, North Carolina
  - San Antonio Military Medical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington
- British Army Training Unit Kenya, Nanyuki, Kenya